CLINICAL TRIAL: NCT04880226
Title: Evaluation of Non Significant Risk Operation Magnetic Resonance Imaging for MR Guided Ablation Using the Philips MRI
Brief Title: A Study to Evaluate Non-significant Risk Operation Magnetic Resonance Imaging for MRI Guided Ablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aiming Lu, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-010671
Record Dates: First submitted 2021-05-06; First posted 2021-05-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: MRI-guided biopsy and/or ablation procedure
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Healthy Volunteers (Other): Imaging of healthy volunteers would performed to optimize image parameters (contrast, SNR) prior to clinical imaging of actual patients receiving treatment.
  Interventions: Device: Magnetic Resonance Imaging (MRI)
- Patients receiving MRI-guided procedures (Experimental): As described in the study protocol this imaging would be performed to evaluate a given sequence for potential benefit during MR-guided interventions.
  Interventions: Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) — Ongoing evaluations of magnetic resonance imaging (MRI) using the Philips Ingenua 1.5T scanner associated with MRI-guided procedures (e.g. ablations or biopsies) are essential to continued procedure improvement within the newly-built hybrid procedure suite.

SUMMARY:
The result of these studies will be used to improve patient care through assessment of new technology to determine whether it is beneficial (i.e. improving data acquisition speed or image quality) during iMRI procedures.

DETAILED DESCRIPTION:
This proposal includes evaluation of advanced MR imaging methods in the iMRI environment and will operate within the NSR guidelines for data acquisition established by the FDA/CDRH. The significant testing by vendor and Mayo staff prior to in vivo use, assure the safety of these studies and overall system stability.

The result of these studies will be used to improve patient care through assessment of new technology to determine whether it is beneficial (i.e. improving data acquisition speed or image quality) during iMRI procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age ≥ 18 years.
* Healthy volunteers or patients already scheduled for a MR-guided procedure.

Exclusion Criteria:

* Individuals 18 years of age.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinical determination whether the sequence improves patient care during MRI-guided procedures. | 3 years
  It will be determined whether the sequence under investigation improves one of the following: 1. lesion targeting (e.g. better guidance of applicators by reduction of metal artifact), 2. lesion ablation (e.g. improved MR thermometry, visualization of cryoablation ice), or 3. accurate assessment of treatment outcome (e.g. margins of ablation relative to lesion boundaries.

CONTACTS AND LOCATIONS:
Overall Officials: Aiming Lu, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States